CLINICAL TRIAL: NCT01234389
Title: Immediate Detection of Helicobacter Infection With a New Electrochemical System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HN-0004
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H. pylori positive patients (Other)
  Interventions: Device: Electrochemical H. pylori detection method; Device: IHC; Device: C13-urea breath test; Device: HUT
- H. pylori negative patients (Other)
  Interventions: Device: Electrochemical H. pylori detection method; Device: IHC; Device: C13-urea breath test; Device: HUT

INTERVENTIONS:
Device: Electrochemical H. pylori detection method — Determination of H. pylori infection.
Device: IHC — Determination of H. pylori infection.
  Other Names: Determination of H. pylori infection.
Device: C13-urea breath test — Determination of H. pylori infection.
Device: HUT — Determination of H. pylori infection.

SUMMARY:
Helicobacter pylori-infection (H. pylori) affects about fifty percent of the general population and is associated with peptic ulcer disease, non-cardia gastric adenocarcinoma and gastric lymphoma. Currently, diagnostic methods include breath tests, serology, stool antigen tests, histology or the Helicobacter urease test (HUT).

The aim of our study is to access the clinical reliability of a new, electrochemical device for rapid H. pylori detection.

DETAILED DESCRIPTION:
The newly developed electrochemical device for H. pylori detection consists of a working and reference electrode between which a biopsy sample is administered. Afterwards, acquired voltage-values could be analysed for characteristics typical for H. pylori infection (ammonia). According to Sydney classification, biopsies are taken from gastric antrum and corpus for electrochemical H. pylori detection, HUT and immunohistochemistry (IHC). HUT results are evaluated after 24 hours. Furthermore, every patient will receive 13C-urea breath test. IHC is designated as the gold standard of H. pylori diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-85 years
* Ability of subjects to understand character and individual consequences of clinical trial
* Subjects undergoing EGD

Exclusion Criteria:

* Inability to provide written informed consent
* Severe Coagulopathy (Prothrombin time < 50% of control, Partial thromboplastin time > 50 s)
* Pregnancy or breast feeding
* Active gastrointestinal bleeding
* Residing in institutions (e.g. prison)
* PPI intake
* antibiotic use, actual or within the last 4 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the newly developed device in comparison to IHC, HUT and C13-urea breath test. | Oktober 2009 - February 2011

CONTACTS AND LOCATIONS:
Overall Officials: Markus F. Neurath, M.D., Ph.D., Study Director — University of Erlangen-Nürnberg; Helmut Neumann, M.D., Ph.D., Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Bavaria, Germany